CLINICAL TRIAL: NCT00147160
Title: Phase II Study of the Combination of Cisplatin + Temozolomide in Malignant Glial Tumours in Children and Adolescents at Diagnosis or in Relapse
Brief Title: Phase II Cisplatin + Temozolomide in Malignant Glial Tumours in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISTEM2; CSET-2002/978
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2006-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide; Cisplatin

INTERVENTIONS:
Drug: Temozolomide, Cisplatinum

SUMMARY:
The purpose of this study is to determine whether the combination of Temozolomide and Cisplatinum is effective in the treatment of malignant glial tumours of children and adolescents

ELIGIBILITY:
Inclusion Criteria:

* Age from 4th birthday and younger than 21st birthday
* Histologically documented malignant glial tumour (WHO classification grade III and IV) : astrocytoma, oligodendroglioma, oligoastrocytoma and mixed tumours
* Measurable and evaluable disease by the imaging criteria (MRI)
* Patient not previously treated by either of the two drugs

Exclusion Criteria:

* Malignant brain stem tumours are excluded

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Estimated)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Radiological response after two courses of Temozolomide-Cisplatinum

SECONDARY OUTCOMES:
Progression-free survival
Health status and quality of life
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Grill, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- Institut Gustave-Roussy, Villejuif, France
- Bristol Royal Hospital for Children, Bristol, United Kingdom